CLINICAL TRIAL: NCT03277105
Title: A Phase 3 Randomized, Multicenter Study of Subcutaneous vs. Intravenous Administration of Daratumumab in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Subcutaneous Versus (vs.) Intravenous Administration of Daratumumab in Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108342; 2017-000206-38 (EudraCT Number); 54767414MMY3012 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Results first posted 2020-07-27 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dara SC (Experimental): Participants will receive a fixed dose of daratumumab as 1800 milligram (mg) subcutaneously (Dara SC) co-formulated with recombinant human hyaluronidase (rHuPH20) 2000 Unit per milliliter (U/mL), once weekly in Cycle 1 and 2, every 2 weeks in Cycle 3 to 6, every 4 weeks in Cycle 7 and thereafter until disease progression, unacceptable toxicity or the end of study. The duration for each cycle is 4 weeks.
  Interventions: Drug: Dara SC
- Dara IV (Active Comparator): Participants will receive daratumumab for intravenous infusion (Dara IV) 16 mg/kg once weekly in Cycle 1 and 2, every 2 weeks in Cycle 3 to 6, every 4 weeks on Day 1 in Cycle 7 and thereafter until disease progression, unacceptable toxicity or the end of study. The duration for each cycle is 4 weeks. For Participants still receiving treatment with Dara-IV at the time of Protocol Amendment 4 the duration of infusion may be shortened to a 90-minute infusion or participants will have the option to switch to Dara 1800 mg subcutaneous (SC) on Day 1 of any cycle, at the discretion of the investigator.
  Interventions: Drug: Dara SC; Drug: Dara IV

INTERVENTIONS:
Drug: Dara SC — Participants will receive a fixed dose of Dara SC as 1800 mg daratumumab with rHuPH20 2000 U/mL, once weekly in Cycle 1 and 2, every 2 weeks in Cycle 3 to 6, every 4 weeks in Cycle 7 and thereafter until disease progression, unacceptable toxicity or the end of study.
Drug: Dara IV — Participants will receive Dara IV 16 mg/kg once weekly in Cycle 1 and 2, every 2 weeks in Cycle 3 to 6, every 4 weeks in Cycle 7 and thereafter until disease progression, unacceptable toxicity or the end of study.
  Other Names: JNJ-54767414
  Arms: Dara IV

SUMMARY:
The purpose of this study is to show that subcutaneous (SC) administration of daratumumab co-formulated with recombinant human hyaluronidase PH20 (Dara SC) is non-inferior to intravenous (IV) administration of daratumumab (Dara IV) in terms of the overall response rate (ORR) and maximum trough concentration (Ctrough).

DETAILED DESCRIPTION:
The study population will consist of adults diagnosed with multiple myeloma who have received at least 3 prior lines of therapy including a proteasome inhibitor (PI) and an immunomodulatory drug (IMiD), or whose disease is refractory to both a PI and an IMiD. The study consists of 3 phases: a screening phase (up to 28 days), a treatment phase, and a follow-up phase. Efficacy, pharmacokinetics, immunogenicity, biomarkers and safety will be assessed at scheduled time. Follow-up will continue until the end of the data collection period, approximately 24 months after the last participant was randomized or when the median overall survival for both arms has been reached, whichever occurs first. The primary hypotheses is that the ORR and maximum Ctrough for Dara SC 1800 milligram (mg) are not inferior to the ORR and maximum Ctrough, respectively, for Dara IV 16 mg per kilogram (mg/kg) in participants with multiple myeloma who have received at least 3 prior lines of therapy including a proteasome inhibitor (PI) and an immunomodulatory drug (IMiD), or whose disease is refractory to both a PI and an IMiD.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a response (Partial response [PR] or better based on investigator's determination of response by international myeloma working group [IMWG] criteria) to at least 1 prior treatment regimen
* Received at least 3 prior lines of therapy including a proteasome inhibitor (PI) (greater than or equal to [>=] 2 cycles or 2 months of treatment) and an immunomodulatory drug (IMiD) (>=2 cycles or 2 months of treatment) in any order during the course of treatment (except for participants who discontinued either of these treatments due to a severe allergic reaction within the first 2 cycles/months). A single line of therapy may consist of 1 or more agents, and may include induction, hematopoietic stem cell transplantation, and maintenance therapy. Radiotherapy, bisphosphonate, or a single short course of corticosteroids (no more than the equivalent of dexamethasone 40 milligram/day [mg/day] for 4 days) would not be considered prior lines of therapy
* Documented multiple myeloma as defined by the criteria below:

  1. Multiple myeloma diagnosis according to the IMWG diagnostic criteria
  2. Measurable disease at Screening as defined by any of the following:

     1. Serum M-protein level >=1.0 gram per deciliter (g/dL) or urine M-protein level >=200 mg/24 hours; or
     2. Light chain multiple myeloma without measurable disease in the serum or the urine: Serum immunoglobulin free light chain (FLC) >=10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Meet the clinical laboratory criteria as specified in the protocol
* Women of childbearing potential must have a negative urine or serum pregnancy test at screening within 14 days prior to randomization

Exclusion Criteria:

* Received daratumumab or other anti-CD38 therapies previously
* Received anti-myeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before the date of randomization. The only exception is emergency use of a short course of corticosteroids (equivalent of dexamethasone 40 mg/day for a maximum of 4 days) before treatment
* Received autologous stem cell transplant within 12 weeks before the date of randomization, or the participant has previously received allogeneic stem cell transplant (regardless of timing)
* Plans to undergo a stem cell transplant prior to progression of disease on this study (these participants should not be enrolled to reduce disease burden prior to transplant)
* History of malignancy (other than multiple myeloma) unless all treatment of that malignancy was completed at least 2 years before consent and the patient has no evidence of disease. Further exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or breast, or other non-invasive lesion, that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (146):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Levine Cancer Institute, Charlotte, North Carolina
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown
  - St Vincents Hospital Melbourne, Fitzroy
  - Alfred Health, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Sir Charles Gairdner Hospital, Nedlands
  - Calvary Mater Newcastle Hospital, Waratah
  - The Queen Elizabeth Hospital, Woodville South
  - Princess Alexandra Hospital, Woolloongabba
- Brazil (11):
  - Fundacao Pio XII, Barretos
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina CEPEN, Florianópolis
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Instituto Joinvilense de Hematologia e Oncologia Ltda Centro de Hematologia e Oncologia, Joinville
  - Associacao Hospitalar Beneficente Sao Vicente de Paulo - Hospital Sao Vicente de Paulo, Passo Fundo
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Instituto de Educacao, Pesquisa e Gestao em Saude, Rio de Janeiro
  - CEHON, Salvador
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Clinica Sao Germano, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - The Gordon & Leslie Diamond Health Care Center, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Victoria Hospital, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHU de Quebec L Hotel Dieu de Quebec, Québec, Quebec
- Czechia (7):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Plzen, Hemato-onkologicke oddeleni, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze - I. interni klinika - klinika hematologie, Prague
- France (7):
  - CHU Caen - Côte de Nacre, Caen
  - Hopital Claude Huriez, Lille
  - CHU de Nantes hotel Dieu, Nantes
  - CHU de Boreaux, Pessac
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
- Alexandra General Hospital of Athens, Athens Attica, Greece
- Israel (7):
  - Hillel Yaffe Medical Center - Oncology, Hadera
  - Rambam Med.Center - Hematology Institute, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Sheba Medical Center Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale Villa Sofia-Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda USL di Piacenza, Piacenza
  - Università di Roma La Sapienza, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - A.O.U. Città della Salute e della Scienza, Torino
- Japan (16):
  - Fukuoka University Hospital, Fukuoka
  - Chugoku Central Hospital, Fukuyama
  - Ogaki Municipal Hospital, Gifu
  - Gunma University Hospital, Gunma
  - Kobe City Medical Center General Hospital, Kobe
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Matsuyama Red Cross Hospital, Matsuyama
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Iwate Medical University Hospital, Numakunai
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka University Hospital, Osaka
  - National Hospital Organization Sendai Medical Center, Sendai
  - National Hospital Organization Shibukawa Medical Center, Shibukawa
  - Japanese Red Cross Medical Center, Shibuya City
- Poland (9):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im Ks B Markiewicza, Brzozów
  - Szpital Uniwersytecki nr 2 im. Jana Biziela w Bydgoszczy, Bydgoszcz
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów
  - Szpitale Pomorskie Sp z o o, Gdynia
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewodzki Szpital Specjalistyczny w Legnicy, Legnica
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im Karola Marcinkowskiego, Poznan
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Russia (11):
  - Emergency Hospital of Dzerzhinsk, Dzerzhinsk
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - City Clinical Hospital # 40, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizny Novgorod
  - Penza Regional Oncology Dispensary, Penza
  - Ryazan Regional Clinical Hospital, Ryazan
  - Saint Petersburg City Hospital #15, Saint Petersburg
  - Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - Samara Region Clinical Hospital, Samara
  - Oncology Dispensary of Komi Republic, Syktyvkar
  - Ekaterinburg City Clinical Hospital # 7, Yekaterinburg
- South Korea (8):
  - Pusan National University Hospital, Busan
  - National Cancer Center, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (13):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Dr. Josep Trueta, Girona
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. de Leon, León
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. de Canarias, San Cristóbal de La Laguna
  - Hosp. Univ. Dr. Peset, Valencia
- Sweden (6):
  - Falu Lasarett, Falun
  - Helsingborgs lasarett, Helsingborg
  - Karolinska University Hospital Huddinge, Huddinge
  - Skanes universitetssjukhus, Lund
  - Norrlands University Hospital, Umeå
  - Akademiska Sjukhuset, Uppsala
- Taiwan (6):
  - Chang-Hua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Ukraine (10):
  - Communal Nonprofit Enterprise 'Cherkasy Regional Oncology Dispensary Of Cherkasy Regional Council', Cherkasy
  - Dnepropetrovsk City Clinical Hospital #4, Regional Hematology Center, Dnipro
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - SI Grigoriev Institute for Medical Radiology National Academy of Medical Science of Ukraine, Kharkiv
  - National Cancer Institute, Dept. of chemotherapy of hemoblastosis, Kiev
  - Kiev Marrow Transplantation Center, Bone Marrow Transplantation Department, Kiev
  - State Institution 'National Scientific Center for Radiation Medicine of NAMS of Ukraine', Kiev
  - Institute of Blood Pathology and Transfusion Medicine of AMS of Ukraine, Lviv
  - Mykolaiv Regional Clinical Hospital, Mykolaiv
  - Ukrainian Medical Stomatological Academy, Poltava Regional Clinical Hospital, Poltava
- United Kingdom (9):
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - Leicester Royal Infirmary - Haematology, Leicester
  - St Bartholomew's Hospital, London
  - Guys St Thomas Hospital, London
  - Christie Hospital NHS Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Royal Marsden Hospital, Surrey
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] LaRoche JK, Lanier J, Alvarenga R, Collins M, Costelloe T, Chiau A, Whetherly H, De Soete W, Faludi J, Rens K. Climate footprint of industry-sponsored in-human clinical trials: life cycle assessments of clinical trials spanning multiple phases and disease areas. BMJ Open. 2025 Feb 19;15(2):e085364. doi: 10.1136/bmjopen-2024-085364. PMID 39971605
- [Derived] Li X, Dosne AG, Perez Ruixo C, Perez Ruixo JJ. Pharmacodynamic-Mediated Drug Disposition (PDMDD) Model of Daratumumab Monotherapy in Patients with Multiple Myeloma. Clin Pharmacokinet. 2023 May;62(5):761-777. doi: 10.1007/s40262-023-01232-8. Epub 2023 Apr 6. PMID 37022569
- [Derived] Usmani SZ, Nahi H, Legiec W, Grosicki S, Vorobyev V, Spicka I, Hungria V, Korenkova S, Bahlis NJ, Flogegard M, Blade J, Moreau P, Kaiser M, Iida S, Laubach J, Magen H, Cavo M, Hulin C, White D, De Stefano V, Lantz K, O'Rourke L, Heuck C, Delioukina M, Qin X, Nnane I, Qi M, Mateos MV. Final analysis of the phase III non-inferiority COLUMBA study of subcutaneous versus intravenous daratumumab in patients with relapsed or refractory multiple myeloma. Haematologica. 2022 Oct 1;107(10):2408-2417. doi: 10.3324/haematol.2021.279459. PMID 35354247
- [Derived] Iida S, Ishikawa T, Min CK, Kim K, Yeh SP, Usmani SZ, Mateos MV, Nahi H, Heuck C, Qin X, Parasrampuria DA, Gries KS, Qi M, Bahlis N, Ito S. Subcutaneous daratumumab in Asian patients with heavily pretreated multiple myeloma: subgroup analyses of the noninferiority, phase 3 COLUMBA study. Ann Hematol. 2021 Apr;100(4):1065-1077. doi: 10.1007/s00277-021-04405-2. Epub 2021 Feb 18. PMID 33599794
- [Derived] Usmani SZ, Mateos MV, Hungria V, Iida S, Bahlis NJ, Nahi H, Magen H, Cavo M, Hulin C, White D, De Stefano V, Fastenau J, Slavcev M, Heuck C, Qin X, Pei H, Masterson T, Lantz K, Gries KS. Greater treatment satisfaction in patients receiving daratumumab subcutaneous vs. intravenous for relapsed or refractory multiple myeloma: COLUMBA clinical trial results. J Cancer Res Clin Oncol. 2021 Feb;147(2):619-631. doi: 10.1007/s00432-020-03365-w. Epub 2020 Aug 27. PMID 32852632
- [Derived] Mateos MV, Nahi H, Legiec W, Grosicki S, Vorobyev V, Spicka I, Hungria V, Korenkova S, Bahlis N, Flogegard M, Blade J, Moreau P, Kaiser M, Iida S, Laubach J, Magen H, Cavo M, Hulin C, White D, De Stefano V, Clemens PL, Masterson T, Lantz K, O'Rourke L, Heuck C, Qin X, Parasrampuria DA, Yuan Z, Xu S, Qi M, Usmani SZ. Subcutaneous versus intravenous daratumumab in patients with relapsed or refractory multiple myeloma (COLUMBA): a multicentre, open-label, non-inferiority, randomised, phase 3 trial. Lancet Haematol. 2020 May;7(5):e370-e380. doi: 10.1016/S2352-3026(20)30070-3. Epub 2020 Mar 23. PMID 32213342

RESULTS

PARTICIPANT FLOW:
Groups:
- Daratumumab IV: Participants received daratumumab intravenous infusion (Dara IV) 16 milligrams per kilogram (mg/kg) once weekly in Cycle 1 and 2, every 2 weeks in Cycle 3 to 6, every 4 weeks thereafter until disease progression, unacceptable toxicity, withdrawal of consent, the investigator decides to stop treatment, or the start of subsequent anticancer therapy. The duration for each cycle was 28 days.
- Daratumumab SC: Participants received daratumumab 1800 mg subcutaneous injection (Dara SC) co-formulated with recombinant human hyaluronidase (rHuPH20) 2000 Units per milliliter (U/mL), once weekly in Cycle 1 and 2, every 2 weeks in Cycle 3 to 6, every 4 weeks thereafter until disease progression, unacceptable toxicity, withdrawal of consent, the investigator decides to stop treatment, or the start of subsequent anticancer therapy. The duration for each cycle was 28 days.
Period: Overall Study
Arm/Group | Daratumumab IV | Daratumumab SC
Started | 259 | 263
Treated (Safety Analysis Set) | 258 | 260
Completed | 0 | 0
Not Completed | 259 | 263
Not completed — Death | 129 | 124
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Other | 118 | 125

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daratumumab IV | Daratumumab SC | Total
Number analyzed (Participants) | 259 | 263 | 522
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (10.16) | 65.3 (9.11) | 66.1 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 127 | 237
  Male | 149 | 136 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 14 | 23
  Not Hispanic or Latino | 227 | 225 | 452
  Unknown or Not Reported | 23 | 24 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 40 | 32 | 72
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 9 | 14
  White | 201 | 207 | 408
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 14 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 15 | 13 | 28
  BRAZIL | 10 | 15 | 25
  CANADA | 16 | 20 | 36
  CZECH REPUBLIC | 20 | 16 | 36
  FRANCE | 6 | 10 | 16
  GREECE | 1 | 6 | 7
  ISRAEL | 5 | 8 | 13
  ITALY | 10 | 16 | 26
  JAPAN | 24 | 18 | 42
  POLAND | 39 | 26 | 65
  RUSSIAN FEDERATION | 28 | 27 | 55
  SOUTH KOREA | 7 | 4 | 11
  SPAIN | 14 | 12 | 26
  SWEDEN | 18 | 18 | 36
  TAIWAN | 6 | 8 | 14
  UKRAINE | 22 | 25 | 47
  UNITED KINGDOM | 16 | 17 | 33
  UNITED STATES | 2 | 4 | 6
Stage of Disease (ISS) [Count of Participants; unit: Participants] — Measure Description: The International Staging System (ISS) consists of following 3 stages - Stage I: serum beta2-microglobulin less than (<) 3.5 milligrams per liter (mg/L) and albumin greater than or equal to (>=) 3.5 grams (g) per 100 milliliter; Stage II: neither stage I nor stage III and Stage III: serum beta2-microglobulin >= 5.5 mg/L.
  Participants
    Stage I | 94 | 82 | 176
    Stage II | 89 | 101 | 190
    Stage III | 76 | 79 | 155
    Data missing or Unknown | 0 | 1 | 1
Number of prior lines [Count of Participants; unit: Participants]
  Less than or equal to (<=) 4 Lines | 175 | 174 | 349
  Greater than (>) 4 Lines | 84 | 89 | 173
Refractory status [Count of Participants; unit: Participants]
  Both protease inhibitor (PI) and immunomodulatory drug (IMiD) | 133 | 125 | 258
  IMiD only | 81 | 67 | 148
  None | 26 | 41 | 67
  PI only | 19 | 30 | 49
Weight group [Count of Participants; unit: Participants]
  <=65 | 92 | 94 | 186
  >65 - 85 | 105 | 102 | 207
  >85 | 61 | 66 | 127
  Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved partial response (PR) or better according to International Myeloma Working Group (IMWG) criteria, during or after study treatment. IMWG criteria for PR: greater than or equal to (>=) 50 percent (%) reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to less than (<) 200 milligrams (mg)/24 hours, If the serum and urine M-proteins are not measurable, a decrease of >=50% in the difference between involved and uninvolved free light chain (FLC) levels were required in place of the M-protein criteria, If serum and urine M-protein are not measurable, and serum free light assay was also not measurable, >=50% reduction in bone marrow plasma cells (PCs) was required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas was also required.
Time Frame: Up to 1 year 8 months
Population: Intent-to-treat (ITT) population included all the randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 259 | 263
Percentage of participants | 39.4 [33.4 to 45.6] | 43.3 [37.3 to 49.6]

2. Primary Outcome: Maximum Trough Concentration (Ctrough) of Daratumumab
Description: Maximum Ctrough was defined as the serum predose concentration of daratumumab on Cycle 3 Day 1.
Time Frame: Predose on Cycle 3 Day 1 (each cycle of 28 days)
Population: Pharmacokinetics (PK) population included participants who received at least 1 administration of study drug and had at least 1 PK sample concentration value after the first dose administration. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 150 | 157
micrograms per milliliter (mcg/mL) | 525 (227) | 611 (318)

3. Secondary Outcome: Percentage of Participants With Treatment-emergent Infusion-related Reactions (IRR)
Description: Percentage of participants with treatment-emergent infusion-related reactions were reported.
Time Frame: Up to 3 years
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 258 | 260
Percentage of participants | 34.5 [28.7 to 40.6] | 12.7 [8.9 to 17.4]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from date of randomization to either progression of disease (PD), death due to any cause, whichever occurs first. IMWG criteria for PD: Increase of 25% from lowest response value in any one of the following: Serum M component (absolute increase must be >=0.5 gram per deciliter (g/dL), Urine M-component (absolute increase must be >=200 mg/24 hours), Participants without measurable serum and urine Mprotein levels: difference between involved and uninvolved free light chain (FLC) levels (absolute increase must be >10 milligrams per deciliter (mg/dL), participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow PC% (absolute percentage must be >=10%), definite development of new bone lesions or soft tissue plasmacytomas or increase in size of bone lesions or tissue plasmacytomas and development of hypercalcemia (serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: Up to 3 years
Population: ITT population included all the randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 259 | 263
Months | 6.08 [4.73 to 7.43] | 5.62 [4.70 to 7.49]

5. Secondary Outcome: Percentage of Participants With Very Good Partial Response (VGPR) or Better
Description: VGPR or better was defined as the percentage of participants who achieved VGPR or better (VGPR, complete response (CR) or stringent complete response [sCR]), based on computerized algorithm as per IMWG criteria during or after the study treatment. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or >=90 percent (%) reduction in serum M-protein plus urine M-protein <100 milligrams (mg)/24 hours, CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells (PCs) in bone marrow. sCR: CR plus normal FLC ratio, and absence of clonal PCs by immunohistochemistry (IHC), immunofluorescencea or 2- to 4 color flow cytometry.
Time Frame: Up to 3 years
Population: ITT population included all the randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 259 | 263
Percentage of participants | 21.6 [16.8 to 27.1] | 23.6 [18.6 to 29.2]

6. Secondary Outcome: Percentage of Participants With Complete Response (Including sCR) or Better
Description: CR or better was defined as percentage of participants with a CR or better (CR or stringent complete response [sCR]) based on computerized algorithm as per IMWG criteria. IMWG criteria for CR- negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow. sCR: CR plus normal FLC ratio, and absence of clonal PCs by IHC, immunofluorescencea or 2- to 4 color flow cytometry.
Time Frame: Up to 3 years
Population: ITT population included all the randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 259 | 263
Percentage of participants | 5.4 [3.0 to 8.9] | 4.6 [2.4 to 7.8]

7. Secondary Outcome: Time to Next Therapy
Description: Time to next therapy was defined as the time from randomization to the start of the first subsequent anti-cancer therapy.
Time Frame: Up to 3 years
Population: ITT population included all the randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 259 | 263
Months | 9.43 [8.15 to 10.71] | 8.80 [7.59 to 10.91]

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of the participant's death due to any cause.
Time Frame: Up to 3 years
Population: ITT population included all the randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 259 | 263
Months | 25.56 [22.05 to NA] — Lower limit of 95% CI were not estimable due to insufficient number of events. | 28.19 [22.77 to NA] — Lower limit of 95% CI were not estimable due to insufficient number of events.

9. Secondary Outcome: Patient-Reported Satisfaction With Therapy as Assessed With Cancer Therapy Satisfaction Questionnaire (CTSQ)
Description: Modified-CTSQ contain 9 items (2 items for Thoughts about Cancer Therapy and 7 items in a defined domain of Satisfaction with Therapy) specific to satisfaction with therapy and for comparison of SC and IV administration. Satisfaction with therapy was calculated based on 7-items using 5-point verbal rating scale, where 1= never and 5= always. Scores were averaged and transformed to a 0-100 scale; higher scores represent better health. At least 5 of the 7 items within the Satisfaction with Therapy domain had to be completed to calculate a domain score. No domain score was calculated for Thoughts about Cancer Therapy.
Time Frame: Cycle 1 (Days 8,15 and 22), Cycle 2 (Days 1,8,15 and 22), Cycle 3,4,5,6,7,8,9,10,11,12,13,14,15,16,17,18,19,20,21 and 22 (Day 1)
Population: ITT population included all the randomized participants. Here, 'N' (number of participants analysed) signifies participants who were evaluable for this outcome measure and 'n' (number of participants analyzed) signifies the number of participants analyzed at a specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 239 | 263
Units on a scale
  Cycle 1 Day 8: number analyzed (Participants) | 227 | 230
  Cycle 1 Day 8 | 70.5 (15.98) | 76.9 (14.64)
  Cycle 1 Day 15: number analyzed (Participants) | 226 | 238
  Cycle 1 Day 15 | 72.1 (16.72) | 78.8 (14.95)
  Cycle 1 Day 22: number analyzed (Participants) | 226 | 239
  Cycle 1 Day 22 | 72.8 (16.20) | 78.7 (15.75)
  Cycle 2 Day 1: number analyzed (Participants) | 239 | 238
  Cycle 2 Day 1 | 74.2 (16.44) | 79.7 (16.58)
  Cycle 2 Day 8: number analyzed (Participants) | 227 | 232
  Cycle 2 Day 8 | 74.8 (15.57) | 80.1 (17.24)
  Cycle 2 Day 15: number analyzed (Participants) | 228 | 224
  Cycle 2 Day 15 | 74.3 (16.94) | 80.0 (17.37)
  Cycle 2 Day 22: number analyzed (Participants) | 221 | 214
  Cycle 2 Day 22 | 75.2 (16.47) | 79.3 (18.65)
  Cycle 3 Day 1: number analyzed (Participants) | 217 | 224
  Cycle 3 Day 1 | 76.0 (17.39) | 80.4 (17.78)
  Cycle 4 Day 1: number analyzed (Participants) | 205 | 209
  Cycle 4 Day 1 | 76.6 (17.22) | 79.5 (19.88)
  Cycle 5 Day 1: number analyzed (Participants) | 187 | 188
  Cycle 5 Day 1 | 77.1 (17.11) | 79.6 (18.95)
  Cycle 6 Day 1: number analyzed (Participants) | 169 | 159
  Cycle 6 Day 1 | 76.1 (17.79) | 81.9 (18.34)
  Cycle 7 Day 1: number analyzed (Participants) | 150 | 137
  Cycle 7 Day 1 | 78.6 (16.01) | 85.0 (16.87)
  Cycle 8 Day 1: number analyzed (Participants) | 135 | 127
  Cycle 8 Day 1 | 79.2 (15.54) | 85.0 (15.18)
  Cycle 9 Day 1: number analyzed (Participants) | 121 | 113
  Cycle 9 Day 1 | 79.8 (15.27) | 85.2 (15.03)
  Cycle 10 Day 1: number analyzed (Participants) | 111 | 103
  Cycle 10 Day 1 | 79.4 (14.73) | 85.8 (13.31)
  Cycle 11 Day 1: number analyzed (Participants) | 96 | 94
  Cycle 11 Day 1 | 79.1 (15.55) | 84.8 (13.50)
  Cycle 12 Day 1: number analyzed (Participants) | 83 | 81
  Cycle 12 Day 1 | 80.3 (15.88) | 85.4 (14.70)
  Cycle 13 Day 1: number analyzed (Participants) | 77 | 76
  Cycle 13 Day 1 | 79.6 (16.57) | 84.4 (15.09)
  Cycle 14 Day 1: number analyzed (Participants) | 60 | 61
  Cycle 14 Day 1 | 80.6 (14.62) | 83.5 (15.54)
  Cycle 15 Day 1: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 1 | 80.2 (15.22) | 86.2 (13.51)
  Cycle 16 Day 1: number analyzed (Participants) | 29 | 29
  Cycle 16 Day 1 | 79.4 (14.84) | 88.5 (13.10)
  Cycle 17 Day 1: number analyzed (Participants) | 15 | 20
  Cycle 17 Day 1 | 79.0 (14.34) | 90.9 (11.26)
  Cycle 18 Day 1: number analyzed (Participants) | 8 | 10
  Cycle 18 Day 1 | 84.8 (14.13) | 91.4 (11.57)
  Cycle 19 Day 1: number analyzed (Participants) | 2 | 8
  Cycle 19 Day 1 | 92.9 (10.10) | 89.3 (13.36)
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 4
  Cycle 20 Day 1 |  | 86.6 (18.53)
  Cycle 21 Day 1: number analyzed (Participants) | 0 | 3
  Cycle 21 Day 1 |  | 84.5 (20.93)
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 22 Day 1 |  | 96.4

10. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the duration from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease according to the IMWG criteria. PD was defined as an increase of 25 % from the lowest response value in one of the following: serum and urine M-component (absolute increase must be >= 0.5 g/dL and >=200 mg/24 hours respectively); Only in participants without measurable serum and urine M-protein levels the difference between involved and uninvolved FLC levels (absolute increase must be > 10 mg/dL); Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: Up to 3 years
Population: Participants analyzed included responders (PR or better) in ITT analysis set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 103 | 115
Months | 10.64 [9.23 to 15.64] | 10.15 [9.23 to 13.77]

11. Secondary Outcome: Time to Partial Response (PR) or Better
Description: Time to PR or better was defined as the time from randomization until onset of first response of PR or better.
Time Frame: Up to 3 years
Population: Participants analyzed included responders (PR or better) in ITT analysis set.
Measure: Median (Full Range); unit: Months
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 103 | 115
Months | 1.02 [0.9 to 24.8] | 1.02 [0.9 to 9.4]

12. Secondary Outcome: Time to Very Good Partial Response (VGPR) or Better
Description: Time to VGPR or better was defined as the time from randomization until onset of first VGPR or better.
Time Frame: Up to 3 years
Population: Participants analyzed included responders (VGPR or better) in ITT analysis set. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 56 | 62
Months | 1.92 [0.9 to 22.8] | 1.95 [1.0 to 19.4]

13. Secondary Outcome: Time to Complete Response (CR) or Better
Description: Time to CR or better was defined as the time from randomization until onset of first CR or better.
Time Frame: Up to 3 years
Population: Participants analyzed included responders (CR or better) in ITT analysis set. Here, 'N' (number of participants analysed) signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Daratumumab IV | Daratumumab SC
Number analyzed (Participants) | 14 | 12
months | 7.23 [1.1 to 14.9] | 9.26 [1.2 to 23.1]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Daratumumab IV | Daratumumab SC
All-Cause Mortality (participants affected / at risk) | 130/258 | 126/260
Serious Adverse Events (participants affected / at risk) | 89/258 | 83/260
Other Adverse Events (participants affected / at risk) | 216/258 | 217/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab IV (N=258) | Daratumumab SC (N=260)
Anaemia (Blood and lymphatic system disorders) | 4 | 6
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Hyperviscosity Syndrome (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular Block (Cardiac disorders) | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 1
Cardiac Failure Chronic (Cardiac disorders) | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Deafness Neurosensory (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 2
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 1 | 2
Chest Discomfort (General disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
General Physical Health Deterioration (General disorders) | 6 | 4
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1
Performance Status Decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Acute Hepatitis B (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Campylobacter Gastroenteritis (Infections and infestations) | 1 | 0
Corona Virus Infection (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 1 | 0
Escherichia Infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Hepatitis B Reactivation (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 3
Listeriosis (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 4 | 3
Lung Infection (Infections and infestations) | 2 | 5
Mastoiditis (Infections and infestations) | 1 | 0
Meningitis Cryptococcal (Infections and infestations) | 0 | 1
Meningitis Pneumococcal (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 13 | 12
Respiratory Syncytial Virus Bronchitis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 2
Rhinovirus Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 4
Septic Shock (Infections and infestations) | 4 | 3
Staphylococcal Sepsis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 2
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood Pressure Increased (Investigations) | 1 | 0
General Physical Condition Abnormal (Investigations) | 0 | 1
Oxygen Saturation Decreased (Investigations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myofascial Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain Oedema (Nervous system disorders) | 1 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Cerebrovascular Insufficiency (Nervous system disorders) | 0 | 1
Iiird Nerve Paralysis (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 1
Confusional State (Psychiatric disorders) | 2 | 0
Acute Kidney Injury (Renal and urinary disorders) | 4 | 4
Haematuria (Renal and urinary disorders) | 0 | 2
Myeloma Cast Nephropathy (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 3
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Circulatory Collapse (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab IV (N=258) | Daratumumab SC (N=260)
Anaemia (Blood and lymphatic system disorders) | 64 | 71
Leukopenia (Blood and lymphatic system disorders) | 10 | 18
Lymphopenia (Blood and lymphatic system disorders) | 17 | 21
Neutropenia (Blood and lymphatic system disorders) | 34 | 52
Thrombocytopenia (Blood and lymphatic system disorders) | 50 | 49
Constipation (Gastrointestinal disorders) | 22 | 16
Diarrhoea (Gastrointestinal disorders) | 32 | 41
Nausea (Gastrointestinal disorders) | 31 | 24
Vomiting (Gastrointestinal disorders) | 21 | 16
Asthenia (General disorders) | 17 | 15
Chills (General disorders) | 32 | 15
Fatigue (General disorders) | 26 | 33
Oedema Peripheral (General disorders) | 15 | 10
Pyrexia (General disorders) | 34 | 36
Bronchitis (Infections and infestations) | 9 | 14
Nasopharyngitis (Infections and infestations) | 21 | 28
Upper Respiratory Tract Infection (Infections and infestations) | 30 | 44
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 33
Back Pain (Musculoskeletal and connective tissue disorders) | 36 | 31
Bone Pain (Musculoskeletal and connective tissue disorders) | 10 | 17
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 16 | 19
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 13 | 15
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 13 | 19
Dizziness (Nervous system disorders) | 11 | 15
Headache (Nervous system disorders) | 25 | 15
Insomnia (Psychiatric disorders) | 14 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 15
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 13 | 10
Hypertension (Vascular disorders) | 23 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03277105/Prot_002.pdf
  • Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT03277105/SAP_001.pdf